CLINICAL TRIAL: NCT03855371
Title: Combination of Decitabine and ATO to Treat AML/MDS Expressing a Classified Type of Mutant p53
Brief Title: Mutant p53-based Personalized Trial Using Decitabine and Arsenic Trioxide on AML/MDS
Acronym: PANDA-T0
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Min Lu, Professor, Ph.D., Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Mutant p53-based trial
Record Dates: First submitted 2017-12-27; First posted 2019-02-26 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: P53 Mutation; Myeloid Malignancy; MDS; Aml
Keywords: p53 mutation; personalized treatment; Decitabine; Arsenic Trioxide; AML; MDS
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Decitabine; Arsenic Trioxide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Decitabine plus arsenic trioxide (Experimental): decitabine: 20mg/m2/d, intravenously, d1-d5, q4w arsenic trioxide: 0.16mg/kg/d, intravenously, d1-d5, q4w(maximum dose: 10mg/d)
  Interventions: Drug: Decitabine; Drug: Arsenic Trioxide

INTERVENTIONS:
Drug: Decitabine — 20mg/m2/d, intravenously, d1-d5, q4w
  Other Names: DAC
Drug: Arsenic Trioxide — 0.16mg/kg/d, intravenously, d1-d5, q4w(maximum dose: 10mg/d)
  Other Names: ATO

SUMMARY:
TP53 mutation is commonly associated with poor cancer patient prognosis yet no mutant p53 (mp53)-targeting regimen was clinically established. Here the investigators try to evaluate the side effect and treatment potential of DAC+ATO in p53 mutated high-risk AML/MDS patients.

About 200 AML/MDS patients will be sequenced for TP53 sequence before recruitment. The investigators estimated about 5 patients, based on the reported p53 mutation frequency in AML/MDS, will be p53-mutated. In the trial, the investigators will selectively recruit the mp53 AML/MDS patients that are predicted to respond to DAC+ATO regimen with highest chance (based on the relevant basic studies).

The investigators designate mutant p53-based clinical trials as 'PANDA (P53 AND Arsenic)-Trials'.

DETAILED DESCRIPTION:
TP53 mutation is commonly associated with poor cancer patient prognosis yet no mutant p53 (mp53)-targeting regimen was clinically established. In two independent clinical trials reported recently, DNA demethylating drug Decitabine (DAC) treatment yielded a surprisingly high rate of complete remission (CR) in mp53-expressing myelodysplastic syndromes (MDS) patients and acute myeloid leukemia (AML) patients. Notably, all of the mp53-expressing patients in the two clinical studies, despite of CR, relapsed quickly. This was attributed to a failure in thoroughly clearing all leukemia-specific mutations and the preexisting mp53 subclone outgrew in all of the relapse patients. Indeed, The investigators also found p53 dysfunctional cells quickly develop a DAC resistance mechanism in cultured tissue (unpublished data). Meanwhile, the investigators found arsenic trioxide (ATO) selectively inhibit p53-mutated cells involving mutant p53 reactivation and mutant p53 degradation (presumably mediated by upregulated mdm2 and RCHY1/Pirh2 through reactivated mutant p53). In addition, DAC and ATO show synergy in inhibiting p53-mutated cells.

In current phase I trial, the investigators try to evaluate the side effect and treatment potential of DAC+ATO in p53 mutated high-risk MDS patients. About 200 AML/MDS patients will be recruited for TP53 sequencing before being trialed. The investigators estimated about 50 patients, based on p53 mutation frequency in AML/MDS, will be sequenced to be mp53-positive. The mp53-positive AML/MDS patients are known to have an extremely poor prognosis. The investigators will select high-risk mp53 MDS patients that are predicted to respond to DAC+ATO with highest chance based on our relevant basic studies.

The other participants (free of p53 mutation) will be excluded from the trial.

ELIGIBILITY:
Inclusion Criteria:

* Occurrence of p53 mutants that are predicted to respond to ATO+DAC with highest chance
* Patients newly diagnosed with myelodysplastic syndromes.
* ECOG Performance status ≤ 3.
* Aged from 18 to 75.
* Active bone marrow hyperplasia indicated by morphology
* Normal liver and renal function, bilirubin ≤35μmol/L, ASL/ALT lower than 2xULN, creatinine level ≤150μmol/L
* Normal cardiac function
* Written Informed consent.

Exclusion Criteria:

* Patients previously treated.
* Confirmed CNS involvement.
* Abnormal liver function which does not meet the inclusion criteria.
* Severe cardiac diseases including myocardial infarction or heart insufficiency.
* QT interval ≥450ms on ECG.
* With other visceral malignancy.
* Active tuberculosis or HIV(+).
* Patients with pregnancy or lactation.
* Allergic or significantly contraindicated to any drugs involved in intervention.
* Significantly contraindicated to HMA chemotherapy.
* ECOG performance status ≥3, CCI >1, ADL <100.
* Unable to understand or follow the study protocol.
* Previous intolerance or allergy history to similar drugs.
* Aged <18 yrs or >75yrs
* MDS patients previously treated with decitabine.
* Participation at same time in another study in which investigational drugs are used.
* Any other conditions interfering the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2018-01-10 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
side effect | during the whole treatment
  evaluate the side effects of current regimen

SECONDARY OUTCOMES:
Overall response rate | at the end of cycle 4 (each cycle is 28 days)
  Partial response (PR) + complete response (CR) rate

CONTACTS AND LOCATIONS:
Overall Officials: Sujiang Zhang, MD, PhD, Principal Investigator — Shanghai Institute of Hematology, Ruijin Hospital
Locations (1):
- Hematological department, Shanghai Institute of Hematology, Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided